CLINICAL TRIAL: NCT05768217
Title: Community Resiliency Collective Efficacy Intervention (CRCEI) for Prevention of Community Violence - A Cluster Randomized Controlled Trial
Brief Title: Community Resiliency Collective Efficacy Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Miller, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22100193; U01CE003524-01 (NIH)
Record Dates: First submitted 2023-02-18; First posted 2023-03-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Violence, Physical; Violence, Non-accidental; Violence, Sexual; Violence, Domestic; Violence, Structural; Violence in Adolescence; Community Violence; Social Cohesion
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: This 2-armed cluster-randomized-controlled community-partnered project will examine the effectiveness of a community-centered intervention that promotes thriving and resiliency to reduce community violence, Community Resiliency Collective Efficacy Intervention (CRCEI). The comparison intervention will be health education sessions, which will occur monthly as a 'light touch' intervention in control neighborhoods to recruit a similar number of community members as in the intervention neighborhoods. The study will be located in Allegheny County in Pennsylvania across 20 neighborhoods (i.e., clusters), such that assigned intervention neighborhoods (n=4) will be matched to similar comparison neighborhoods (n=4), and 12 neighborhoods will be randomized either to receive the Collective Efficacy program (i.e., intervention neighborhood, n=6) or to health sessions (comparison neighborhood, n=6). Community surveys will examine neighborhood perspectives before and after program implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Resiliency Collective Efficacy Intervention (CRCEI) (Experimental): Community Resiliency Collective Efficacy Intervention (CRCEI) to engage community members in dialogue on thriving, community leadership, and organizing for social change (9 sessions).
  Interventions: Behavioral: Community Resiliency Collective Efficacy Intervention (CRCEI)
- Health Education Sessions (Active Comparator): Comparison neighborhoods will receive health education sessions as a control intervention. (9 sessions)
  Interventions: Behavioral: Health Education Sessions

INTERVENTIONS:
Behavioral: Community Resiliency Collective Efficacy Intervention (CRCEI) — The Community Resiliency Collective Efficacy Intervention (CRCEI) will involve community members in dialogue on thriving, community leadership, and organizing for social change. Participants in the intervention condition will be asked to participate in 2 sessions of discussions about community thriving and a 7-week training program on the following topics: Building on the Strengths of Your Community, Collective Efficacy and its Effects on Violence Prevention & Community Mental Health, Non-threatening Peaceful Intervention Principles and Strategies: Part One, Non-threatening Peaceful Intervention Principles and Strategies: Part Two, Safety and Roles of Police and Community in Intervening, Active/Effective listening and non-violent communication skills, and Community Resources and Indirect Intervention.
  Arms: Community Resiliency Collective Efficacy Intervention (CRCEI)
Behavioral: Health Education Sessions — Comparison neighborhoods will receive health education sessions across a variety of community-identified health topics as a control intervention. (9 sessions)
  Arms: Health Education Sessions

SUMMARY:
This study will evaluate, via a cluster-randomized controlled trial, the effectiveness of a community-centered intervention that promotes thriving and resiliency to reduce community violence.

DETAILED DESCRIPTION:
This study will evaluate, via a cluster-randomized controlled trial, the effectiveness of an innovative community-centered intervention that promotes thriving and resiliency to reduce community violence. In collaboration with community partners, this study will implement a Community Resiliency Collective Efficacy Intervention (CRCEI) to engage community members in dialogue on neighborhood transformation, racial and gender equity, community leadership, and organizing for social change. Facilitating discussion and community organizing within neighborhoods about child and youth thriving is expected to increase individual and neighborhood levels of collective efficacy and reduce community violence. Using a community-partnered participatory approach, this study will use a Community Thriving Matrix tool to engage youth and adult community members in ongoing dialogue on neighborhood transformation, community leadership, and organizing for social change. This focus on envisioning and creating neighborhoods in which children and adolescents can thrive is expected to translate to increased individual and neighborhood levels of collective efficacy as well as violence reduction. Comparison neighborhoods will receive health education sessions as a control intervention. The proposed study involves diverse neighborhoods in the Pittsburgh region and collecting survey data from youth (ages 13-19 years) and adult community participants (both male and female identified). Interviews with a sub-sample of community residents and facilitators and community site leads as well as observations of intervention delivery will provide qualitative information on processes of program implementation. This study will provide the first rigorous evaluation of this community-level prevention approach.

ELIGIBILITY:
Inclusion Criteria:

* youth age 13 years old and up (all genders)
* adults 18 years and older (all genders)
* reside in neighborhoods selected to participate in the study

Exclusion Criteria:

* individuals younger than 13 years old

  * individuals residing outside of participating neighborhoods

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4600 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in perceptions of neighborhood collective efficacy and community cohesion | Change from baseline to approximately 12 months after baseline
  Composite Measure mean score (range 1 - 5; 1 is low and 5 is best) of neighborhood-level perceptions of collective efficacy and community cohesion

SECONDARY OUTCOMES:
Community incidence of violence in 12 month period | Change from 1 year period before baseline to approximately 12 months after baseline
  number of incidents of violence, i.e., assaults, gun violence, referrals to child protective services, compared to control neighborhoods.
Community incidence of violence in 12 month period | Change from 1 year period before baseline to approximately 2 years after baseline
  number of incidents of violence, i.e., assaults, gun violence, referrals to child protective services, compared to control neighborhoods.
Change from baseline in collective efficacy and neighborhood social norms | Change from baseline to approximately 12 months after baseline
  Composite Collective Efficacy Measure mean score (range 1-5; 1 is lowest and 5 is best) of individual-level collective efficacy and neighborhood social norms
Number of self-reported events of violence exposure | Change from baseline to approximately 12 months after baseline
  count of individual-level events of violence exposure

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We do not plan to make a fully documented, publicly available data set on a website for download because while individual participant data are de-identified, it could be possible to discern the neighborhoods or sites from the dataset and therefore compromise the anonymity of the data. Therefore, we will make the data available only to selected researchers who apply for access. The application must document a legitimate public health use or research question for the data, and the applicant must sign a pledge to keep all data private and to make no attempt to identify individual subjects. This use of the data is consistent with the planned language of the voluntary consent for participation agreed and in accordance with IRB policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after data collection is completed.
Access Criteria: Data sharing agreement must be completed with investigators and the University of Pittsburgh.